CLINICAL TRIAL: NCT04785833
Title: A Prospective, Open, Single-arm Clinical Study on the Efficacy and Safety of CD7 CAR-T in the Treatment of CD7-positive Refractory Relapsed Acute Leukemia
Brief Title: CD7 CAR-T in the Treatment of CD7 Positive Refractory Relapsed Acute Leukemia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: PersonGen BioTherapeutics (Suzhou) Co., Ltd. (Industry)
Collaborators: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PA-CART-3-17-001
Record Dates: First submitted 2021-03-03; First posted 2021-03-08 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2021-03

CONDITIONS: T-ALL
MeSH Terms: conditions — Precursor T-Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- T cell injection targeting CD7 chimeric antigen receptor (Experimental)
  Interventions: Drug: T cell injection targeting CD7 chimeric antigen receptor

INTERVENTIONS:
Drug: T cell injection targeting CD7 chimeric antigen receptor — Drug name: T cell injection targeting CD7 autologous chimeric antigen receptor. Package specification: 10-50ml bag, 1-4 bags / person, which is determined according to the body weight of the subject and the effective content of cell preparation

SUMMARY:
Patients with acute leukemia derived from T lymphocytes have the characteristics of high expression of CD7 antigen, such as acute T lymphocyte leukemia (T-ALL).CAR-T therapy is to genetically modify the patient's T lymphocytes to target and eliminate tumor cells in a major histocompatibility complex-independent manner. CAR-T cells are costimulatory molecules that include single-chain antibodies (scFv) that recognize tumor-specific antigens, hinge regions, transmembrane regions, intracellular signaling regions (immunoreceptor tyrosine activation motif ITAM), and intracellular signaling regions. The chimeric antigen receptor of CD28 or CD137(4-1BB) conduction domain is expressed in a lentiviral vector, and the vector is transfected into autologous T cells, so that the modified CAR-T cells have targeting and specificity Recognizes and kills cancer cells expressing tumor antigens, and can proliferate and activate in vivo, but has no effect on cells that do not express the antigen

ELIGIBILITY:
Inclusion Criteria:

* Age 12-65
* Sign informed consent
* Expected survival time ≥ 3 months
* CD7 positive refractory and relapsed acute leukemia
* Karnofsky score≥60
* ECOG score ≤ 2
* Have not received other immunotherapy within 3 months
* The CD7 expression rate on the surface of leukemia cells detected by flow cytometry is greater than 30%

Exclusion Criteria:

* Uncontrolled active infection
* Active viral hepatitis B or C
* HIV test positive
* Congenital immunodeficiency patients
* Pregnant and breastfeeding patients
* Patients with central nervous system tumors or central nervous system leukemia
* The patient and/or family members do not agree to the treatment plan

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-03-04 (Estimated); Primary Completion 2022-04-30 (Estimated); Study Completion 2024-02-04 (Estimated)

PRIMARY OUTCOMES:
DLT | Up to 2 years
  Dose-limiting toxicity

SECONDARY OUTCOMES:
Safety results | Up to 2 years
  Number of adverse events
PK | Up to 2 years
  The maximum concentration (Cmax）
PD | Up to 2 years
  Absolute value of CD7 Positive Cells in peripheral blood at each time point

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliared Hospital Of SOOCHOW University, Suzhou, Jiangsu, China